CLINICAL TRIAL: NCT05590312
Title: Comparison of Changes in Total Oxidant and Total Antioxidant Capacities in Low-Flow and High-Flow General Anesthesia Protocols
Brief Title: Comparison of Total Oxidant and Total Antioxidant Capacities in Low-Flow and High-Flow General Anesthesia
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Özlem Ersoy Karka, Assistant Professor, Duzce University
Other Study IDs: drozlemersoy3
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Oxidative Stress; Anesthesia
Keywords: Oxidative stress; Anesthesia, General; Low flow anesthesia
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low Flow Group - Group D: Vitamin D, Albumin, CRP, TAS and TOS values will be checked before and during the operation in 36 patients who will receive general anesthesia. Flow of 1 L/min will be given during the operation. The processed EEG values of all patients will be monitored and they will be ensured to be at the same anesthesia depth. Albumin, CRP, TAS and TOS values will be checked again from the blood taken postoperatively in the patients who were taken to the service after the operation and these values will be compared with the previous ones.
  Interventions: Other: general anesthesia
- High Flow Group - Group Y: Vitamin D, Albumin, CRP, TAS and TOS values will be checked before and during the operation in 36 patients who will receive general anesthesia. Flow of 4 L/min will be given during the operation. The processed EEG values of all patients will be monitored and they will be ensured to be at the same anesthesia depth. Albumin, CRP, TAS and TOS values will be checked again from the blood taken postoperatively in the patients who were taken to the service after the operation and these values will be compared with the previous ones.
  Interventions: Other: general anesthesia

INTERVENTIONS:
Other: general anesthesia — All patients will undergo general anesthesia. Group D will receive fresh gas flow of 1 l/min and Group Y will receive fresh gas flow of 4 l/min.

SUMMARY:
The goal of this observational study is to determine whether low-flow anesthesia has a positive contribution to the total oxidant/antioxidant balance.

DETAILED DESCRIPTION:
General anesthesia is a complex physiological state characterized by reversible loss of consciousness, whole-body analgesia, amnesia, and muscle relaxation. Modern anesthesia devices used for patients under general anesthesia are semi-closed rebreathing systems. The fresh gas flow entering these closed systems is determined by the anesthetists.

The term low-flow anesthesia is used to describe inhalation anesthesia techniques that are administered with a semi-closed rebreathing system and have a rebreathing rate of at least 50%. The high standard of anesthesia machines, the existence of monitors that analyze the anesthetic gas composition continuously and in detail, and the increase in knowledge about the pharmacodynamics and pharmacokinetics of inhalation anesthetics have greatly facilitated the safe administration of low-flow anesthesia. The terminology associated with low-flow anesthesia techniques may be based on rebreathing rate or fresh gas flow rate. The most important factor determining the rebreathing rate is the fresh gas flow rate. If the fresh gas flow rate is reduced to less than 2 L/min when using modern rebreathing systems, low-flow anesthesia can be mentioned for most patients.

Oxidative stress is accepted as a pathological mechanism. Oxidative stress is a state of oxidative damage that occurs when the critical balance between free radical production and antioxidant defense systems is disrupted. Oxidative stress is beneficial in certain physiological conditions. For example, it can strengthen biological defense mechanisms during appropriate physical exercise and ischemia. However, its benefits are limited to these specific situations, and in many other cases, high levels of oxidative stress cause cell death and thus cell and tissue damage via necrotic or apoptotic mechanisms. If damage continues at the cell and tissue level, it causes the onset and progression of various organ damage and diseases.

Aim: In low-flow anesthesia applications, the amount of inspired oxygen is expected to be low due to keeping the gas supplied to the system low. Therefore, in this study, it will be investigated whether low-flow anesthesia has a positive contribution to the total oxidant/antioxidant balance.

Method: A total of 72 patients undergoing general anesthesia who meet the inclusion criteria and signed informed consent will be included in the study. Vitamin D, albumin, C-reactive protein (CRP), Total Antioxidant (TAS) and Total Oxidant (TOS) levels will be determined in the blood samples taken from all volunteers routinely before the operation. Basal peak heart rate (HR), peripheral oxygen saturation (SpO2), systolic (SBP) and diastolic blood pressure (DBP), end-tidal carbon dioxide (ETCO2), body temperature and processed EEG values will be recorded. All measurements will be recorded and repeated at 5 minute intervals throughout the operation. Volunteers will be randomly divided into 2 groups as low flow group (D) and high flow group (Y). Fresh gas flow of 1 L/min to D group and 4 L/min to Y group will be administered. During the operation, the processed EEG values of all patients will be held between 40-60 and it will be ensured that they are at the same anesthesia depth. Albumin, CRP, TAS and TOS values will be checked again in the blood samples taken for routine tests performed at the end of operation and postoperatively within 6-24 hours after the end of operation, and these values will be compared with the values obtained before the operation.

Statistical Analysis: It is planned to use 'Independent Samples t test' or 'Mann-Whitney U test' in comparison of the groups, depending on the distribution of the data. Chi-square tests will be used to examine the relationships between categorical variables. 'Repeated Measure ANOVA' will be used in the evaluation of repeated measurements. Correlations between continuous variables will be analyzed by Pearson or Spearman correlation analysis, depending on the distribution of the data.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years and younger than 60 years of age who will be operated under general anesthesia
* Patients in I, II risk groups according to the American Society of Anesthesiologists (ASA) classification

Exclusion Criteria:

* ASA III and above patients,
* Patients for whom Intensive Care Unit (ICU) indication is required
* Chronic obstructive pulmonary disease,
* Personal or family history of malignant hyperthermia,
* Morbid obesity,
* Alcohol or drug dependency,
* Having a history of liver or kidney disease,
* Having coronary artery disease or heart failure,
* Having significant anemia or hemoglobinopathy,
* Hypotension, hypovolemia, sepsis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 72 patients who meet the inclusion criteria and sign informed consent will be included.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Ersoy Karka, Principal Investigator — Düzce University Faculty of Medicine
Locations (1):
- Duzce University Faculty of Medicine, Düzce, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Flow Group - Group D | High Flow Group - Group Y
Started | 36 | 36
Completed | 36 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Flow Group - Group D | High Flow Group - Group Y | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 36 | 72
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (11) | 39 (12) | 37 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 20 | 21 | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 36 | 36 | 72
Fresh gas flow [Number; unit: liter/minute] | 1 | 4 | 2.5

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Total Antioxidant Status (TAS) Levels Between the Two Groups
Description: Vitamin D, Albumin, CRP, TAS and TOS values will be checked before the operation in 72 patients who will receive general anesthesia in both groups. Albumin, CRP, TAS and TOS values will be checked again from the blood taken postoperatively in the patients who were taken to the ward after the operation and these values will be compared between two groups and with the previous level in the same group.
Time Frame: 3 times in 24 hours perioperatively. TAS/TOS levels will be determined before the operation, at the end of operation and at 6th hour after the end of operation.
Measure: Mean (Standard Deviation); unit: mmol Eq / L
Arm/Group | Low Flow Group - Group D | High Flow Group - Group Y
Number analyzed (Participants) | 36 | 36
mmol Eq / L
  T0: Before the operation | 1.76 (0.23) | 1.82 (0.3)
  T1: At the end of the operation | 1.83 (0.24) | 1.92 (0.27)
  T2: At 6th hour after the end of the operation | 1.85 (0.28) | 1.89 (0.29)

2. Primary Outcome: Change From Baseline in Total Oxidant Status (TOS) Levels
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: µmol H2O2 q/L
Arm/Group | Low Flow Group - Group D | High Flow Group - Group Y
Number analyzed (Participants) | 36 | 36
µmol H2O2 q/L
  T0: before the operation | 19.82 (11.82) | 21.48 (11.01)
  T1: at the end of operation | 19.66 (11.75) | 17.20 (8.72)
  T2: at 6th hour after the end of operation. | 22.49 (11.99) | 21.38 (11.64)

3. Primary Outcome: Change From Baseline in Albumin Levels.
Description: as for outcome 1
Time Frame: 3 times in 24 hours perioperatively. Albumin levels will be determined before the operation, at the end of operation and at 6th hour after the end of operation.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Low Flow Group - Group D | High Flow Group - Group Y
Number analyzed (Participants) | 36 | 36
mg/dL
  T0: before the operation | 4.24 (0.3) | 4.15 (0.24)
  T1: at the end of operation | 4.05 (0.38) | 4.02 (0.39)
  T2: at 6th hour after the end of operation. | 3.96 (0.36) | 3.97 (0.40)

4. Primary Outcome: Change From Baseline in C Reactive Protein (CRP) Levels.
Description: as for outcome 1
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Low Flow Group - Group D | High Flow Group - Group Y
Number analyzed (Participants) | 36 | 36
mg/dL
  T0: before the operation | 0.30 (0.54) | 0.53 (1.61)
  T1: at the end of operation | 0.31 (0.56) | 0.52 (1.36)
  T2: at 6th hour after the end of operation. | 1.41 (2.58) | 1.37 (2.31)

5. Primary Outcome: Comparison of Vitamin D Levels Between the Two Groups
Description: as for outcome 1
Time Frame: 1 time before the operation.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Low Flow Group - Group D | High Flow Group - Group Y
Number analyzed (Participants) | 36 | 36
mg/dL | 7.5 (10.9) | 14.8 (13)

ADVERSE EVENTS:
Time Frame: 2 days: operation day and postoperative 6 hours ( postoperative 1st day)
Description: Number of Participants at Risk is equal to the number of participants assigned to both study groups. 72 patients are at risk of adverse events.
Arm/Group | Low Flow Group - Group D | High Flow Group - Group Y
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT05590312/Prot_SAP_000.pdf